CLINICAL TRIAL: NCT06122532
Title: Clinical Study on Umbilical Cord Mesenchymal Stem Cells for Wound Repair in Large Area Burn Patients
Brief Title: Umbilical Cord Mesenchymal Stem Cells for the Repair of Large Area Burn Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShiCang Yu (Other)
Responsible Party: Sponsor-Investigator, ShiCang Yu, Director, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zsyx3
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Large Area Burns
Keywords: Large area burns; human umbilical cord mesenchymal stem cells; wound healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stem cell preparation combined with Reticular skin (Experimental)
  Interventions: Procedure: Stem cell preparation combined with Reticular skin
- Stem cell preparation combined with MEEK skin (Experimental)
  Interventions: Procedure: Stem cell preparation combined with MEEK skin
- Stem cell preparation combined with split-thickness skin (Experimental)
  Interventions: Procedure: Stem cell preparation combined with split-thickness skin
- autologous skin grafting (Placebo Comparator)
  Interventions: Procedure: autologous skin grafting

INTERVENTIONS:
Procedure: Stem cell preparation combined with Reticular skin — The dose of transplanted stem cells per wound (100cm2) is 1×10^6, then cover the wound with autologous regular skin.
  Arms: Stem cell preparation combined with Reticular skin
Procedure: Stem cell preparation combined with MEEK skin — The dose of transplanted stem cells per wound (100cm2) is 1 × 10 ^ 6, then cover the wound with autologous MEEK skin.
  Arms: Stem cell preparation combined with MEEK skin
Procedure: Stem cell preparation combined with split-thickness skin — The dose of transplanted stem cells per wound (100cm2) is 1 × 10 ^ 6, then cover the wound with autologous split-thickness skin.
  Arms: Stem cell preparation combined with split-thickness skin
Procedure: autologous skin grafting — After cleaning the wound, use autologous skin (Reticular skin/MEEK skin/split-thickness skin) grafting and cover the wound surface。
  Arms: autologous skin grafting

SUMMARY:
This study intends to adopt a prospective, open, and randomized controlled research method to explore the effectiveness and safety of using human umbilical cord mesenchymal stem cells to treat large-scale burn wounds, in order to break through the limitations of various current treatment methods, explore new clinical treatment methods, promote the repair and healing of skin lesions, and further improve the cure rate and quality of life of patients.

DETAILED DESCRIPTION:
Large area deep burn patients, due to extensive skin defects in their limbs that cannot be repaired by the body itself, need to undergo skin grafting surgery to seal the wound. Although skin transplantation can partially meet the needs of wound sealing, the skin scar hyperplasia after transplantation and healing is significant, affecting the appearance and motor function of the limbs. Moreover, the healed skin lacks dermal tissue and sweat glands and other skin accessories, resulting in poor skin quality after wound healing, And accompanied by obvious discomfort such as fear of heat, itching, and pain, which seriously affects the patient's quality of life. Mesenchymal stem cells have high differentiation potential and can differentiate across embryonic boundaries into epithelial tissue cells such as skin. They can also secrete various cytokines to produce chemotactic and anti apoptotic effects, promoting the formation of wound neovascularization and wound healing. Human umbilical cord mesenchymal stem cells, due to their convenient and painless source, have become good seed cells for promoting wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients are voluntary and sign an "informed consent form";
2. Burn wound area ≥ 20% TBSA, and III ° wound area ≥ 2% TBSA;
3. Age range from 18 to 65 years old, regardless of gender;
4. Plan to perform two or more limb III degree wounds with scab cutting and autologous skin grafting surgery for treatment;
5. No severe heart, lung, blood system, or nervous system diseases;
6. There are no clear complications such as systemic infections.

Exclusion Criteria:

1. Patients who do not agree to participate in this experimental study;
2. Age<18 years old or>65 years old;
3. Patients with definite malignant tumors, AIDS, diabetes, and autoimmune diseases;
4. Pregnant or lactating patients;
5. Individuals with systemic dysfunction;
6. Patients with acute and chronic liver and kidney diseases;
7. Poor compliance makes it difficult to complete the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate | On the 21st and 28th days after surgery
  (Total area of wound in the operating area - area of unhealed wound)/Total area of wound in the operating area × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Army Medical University (Third Military Medical University), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No